CLINICAL TRIAL: NCT03152981
Title: Analysis of Change of Optic Nerve Sheath Diameter Using Ultrasonography in Robot Assisted Laparoscopic Radical Prostatectomy
Brief Title: Analysis of Change of Optic Nerve Sheath Diameter in Robot Assisted Laparoscopic Radical Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-1602/335-006
Record Dates: First submitted 2017-04-23; First posted 2017-05-15 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2017-05

CONDITIONS: Optic Nerve Sheath Diameter; Robot Assisted Laparoscopic Radical Prostatectomy
MeSH Terms: interventions — Desflurane; Propofol; Remifentanil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Desflurane group (Active Comparator): In desflurane group, desflurane 6-8 vol% and remifentanil (target controlled infusion 2-3 ng / ml) are used for maintenance of anesthesia during surgical procedure
  Interventions: Drug: Desflurane; Drug: remifentanil
- Propofol group (Active Comparator): In propofol group, propofol 3-4 ug/ml and remifentanil 2-3 n /ml using target Controlled Infusion are used for maintenance of anesthesia during surgical procedure
  Interventions: Drug: propofol; Drug: remifentanil

INTERVENTIONS:
Drug: Desflurane — In desflurane group, desflurane 6-8 vol% and remifentanil (target controlled infusion 2-3 ng / ml) are used for maintenance of anesthesia during surgical procedure. In propofol group, propofol 3-4 ug/ml and remifentanil 2-3 n /ml using target Controlled Infusion are used for maintenance of anesthesia during surgical procedure
  Other Names: DES
  Arms: Desflurane group
Drug: propofol — In desflurane group, desflurane 6-8 vol% and remifentanil (target controlled infusion 2-3 ng / ml) are used for maintenance of anesthesia during surgical procedure. In propofol group, propofol 3-4 ug/ml and remifentanil 2-3 n /ml using target Controlled Infusion are used for maintenance of anesthesia during surgical procedure
  Other Names: PPF
  Arms: Propofol group
Drug: remifentanil — In desflurane group, desflurane 6-8 vol% and remifentanil (target controlled infusion 2-3 ng / ml) are used for maintenance of anesthesia during surgical procedure. In propofol group, propofol 3-4 ug/ml and remifentanil 2-3 n /ml using target Controlled Infusion are used for maintenance of anesthesia during surgical procedure
  Other Names: Remi

SUMMARY:
In the present study, The investigators evaluated whether anesthetic agents effects on Optic Nerve Sheath Diameter in patients undergoing Robot Assisted Laparoscopic Radical Prostatectomy

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing robotic laparoscopic radical prostatectomy
2. Adults 20 to 80 years of age
3. American Society of Anesthesiologists Physical grade 1-2

Exclusion Criteria:

1. Patients who did not agree to participate in the study
2. Patients with ophthalmic diseases
3. Patients with previous history of ophthalmic surgery
4. Patients with neurological disorders
5. Patients with history of head surgery due to neurological disorders

Ages: 20 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-06-03 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Optic Nerve Sheath Diameter | 1 hour after Trendelenburg position

CONTACTS AND LOCATIONS:
Overall Officials: Eunsu Choi, Pf, Study Chair — Seoul National Univ. Bundang Hospita
Locations (1):
- Seoul National Univ. Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea